CLINICAL TRIAL: NCT02912611
Title: Detection and Management of Acute Kidney Injury (AKI) in Low and Low Middle Income Countries: A Pilot Feasibility Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: International Society of Nephrology (Other)
Responsible Party: Principal Investigator, Ravindra Mehta, Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 160610
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moderate and High risk for AKI (Other)
  Interventions: Procedure: Education and Protocol based management

INTERVENTIONS:
Procedure: Education and Protocol based management

SUMMARY:
This feasibility study will be conducted at 4 international sites located in Asia (Dhahran, Nepal); Africa (Blantyre, Malawi and Kilimanjaro, Tanzania) and Latin America (Cochabamba, Bolivia).

Each site comprises a cluster (including 3-4 health centers - 1 district hospital - 1 regional referral hospital) that service the population around the site area. Patients presenting at a health care clinic or hospital emergency department with signs and symptoms associated with high and moderate risk of developing AKI will undergo a point of care (POC) test to measure serum creatinine, saliva urea nitrogen dipstick (exclusively in Malawi), and a urine dipstick test for color, protein, glucose, blood and specific gravity. Patients who meet the study inclusion criteria will be approached for consent. Patients enrolled in the study will be followed throughout the health care evaluation and tracked through their course by location i.e. health care center, hospital, and home. Outcomes will be recorded through 6 months following the health care evaluation.

The protocol will have an initial observation phase, during which relevant healthcare staff and the research team will be trained to identify patients at moderate or high risk of AKI and use of the point of care (POC) test for serum creatinine, saliva urea nitrogen dipstick (exclusively in Malawi), and urine dipstick test. During this phase patients will be tracked throughout the health care evaluation, however the teleconsultation will not be implemented and no specific guidance for managing the patient will be provided.

During the subsequent intervention phase, the research team will interact with the local healthcare providers to and the teleconsultation physician, providing guidance on the management of the patient based on a standardized protocol. Protocols for patient care will be pre-specified, with minor adjustments to meet local requirements.

ELIGIBILITY:
Inclusion Criteria:Presence of Signs and Symptoms determining AKI risk

* Decreased urine volume
* Hypotension/ shock
* Coma
* Jaundice
* Confusion
* Dyspnea
* Symptoms of respiratory infection
* Petechia, ecchymosis, bleeding
* Hypertension (in pregnancy)

Exclusion Criteria:

* Chronic kidney disease in patients receiving regular dialysis treatment
* Kidney transplant patients
* Unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2101 (Actual)
Dates: Start 2016-10-01; Primary Completion 2017-09-29 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility of implementing an education and training program to optimize care of AKI | 1 year
  Managment will be based on a protocol driven comprehensive 5R (Risk, Recognition, Response, Renal Support and Rehabilitation) approach in resource constrained regions in Africa, Asia and Latin America.

CONTACTS AND LOCATIONS:
Locations (3):
- Hospital Obrero #2, Cochabamba, Bolivia
- Queen Elizabeth Central Hospital (QECH), Blantyre, Malawi
- BP Koirala Institute of Health Sciences, Dharān, Sansari District, Nepal

IPD SHARING:
Plan to Share IPD: Undecided